CLINICAL TRIAL: NCT06603896
Title: Effects of Single and Combined Aromatherapy on Nursing Student Anxiety, Test Anxiety, Nausea or Queasiness, Exam Grades, GPA, and Perceived Stress
Brief Title: Effects of Different Aroma-therapies on Nursing Students.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pace University (Other)
Responsible Party: Principal Investigator, Martha J.Greenberg, Professor, Pace University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: PaceU
Record Dates: First submitted 2024-09-07; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Nausea; Stress; Anxiety; Aromatherapy
Keywords: aromatherapy; nursingstudent; testanxiety; nausea; GPA; stress
MeSH Terms: conditions — Nausea; Anxiety Disorders | interventions — Aromatherapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo group (Sham Comparator): a sham unscented aromatherapy patch will be applied to subjects clothing, 4-6 inches below the neck on the thorax
  Interventions: Other: Aromatherapy
- Combined Aromatherapy Group (Active Comparator): A combined scents Citrus Lavendar infused aromatherapy patch will be applied to subjects clothing, 4-6 inches below the neck on the thorax
  Interventions: Other: Aromatherapy
- Single Aromatherapy Lavendar Group (Active Comparator): A single scent Lavander aromatherapy patch will be applied 4-6 inches below nose on front of thorax on subjects clothing
  Interventions: Other: Aromatherapy

INTERVENTIONS:
Other: Aromatherapy — Aromatherapy and placebo patches will be used

SUMMARY:
The aim of this study is to investigate the use of lavender and citrus inhalation aromatherapy on anxiety, test anxiety and sleep quality in Pace University sophomore, junior and senior nursing majors. Anxiety, particularly test anxiety, is a ubiquitous problem among nursing students. Test anxiety is a type of state anxiety experienced as concern or fear before, during, or following a test or performance assessment. While some anxiety may enhance the performance of a student, test anxiety often negatively effects performance. Although test anxiety can be incapacitating to any student, in nursing students it can not only have a negative impact on learning, it is a major cause for under-achievement and prevents some students from reaching their academic potential since they are enrolled in a high-stakes program.

Treatment for test anxiety includes counseling, desensitization therapy, relaxation therapies, and aromatherapy. Aromatherapy with its focus on the therapeutic use of plant oils has the ability to decrease anxiety in humans through the use of natural oils particularly Lavandula angustifolia (lavender) without the potential for adverse reactions or side effects of conventional anxiolytic drugs.

Research on the efficacy of aromatherapy on test anxiety in college and nursing students shows mixed results. A variety of designs and essential oil scents, either mixed or single, were used with subjects, e.g., lavender, rosemary, peppermint, lemon and the vehicles used to administer the oils, e.g., room diffused inhalation, non-absorbent cloth infused lavender for the aromatherapy vary.

However, studies using lavender essential oil to reduce anxiety in college students, nursing students, and patients, demonstrated that lavender overall acted as an effective anxiolytic in reducing the stress of test taking, especially with lower levels of anxiety. Thus lavender essential oil could benefit nursing students in reducing test anxiety, and has great potential in benefiting all students in test and anxiety reduction, provided the person is not allergic to the oil. There is support for the notion that aromatherapy is a safe intervention, in a systematic review on the anxiolytic effects of aromatherapy in people with anxiety symptoms, no participants reported experiencing any adverse effects., The use of lavender also appears to help sleep without the adverse effects of commonly used drugs. The anxiolytic effects of the oil might reduce unhealthy behaviors that students engage in, e.g. alcohol and drug use/overuse, to reduce stress and relax, and positively affect sleep. In a 2015-2016 study of Pace nursing students, the results showed improvement in sleep and test anxiety, although the sample was small.

DETAILED DESCRIPTION:
The study will identify subjects test anxiety and poor sleep quality and reduction in anxiety prior to/ during performance assessments as a result of the anxiolytic properties of the lavender essential oil inhaler we will provide them with and potentially improvement in quality of sleep. Studies using lavender essential oil to reduce anxiety in college students, and patients, demonstrated that lavender overall acted as an effective anxiolytic in reducing the stress of test taking, especially with lower levels of anxiety. Thus lavender essential oil could benefit nursing students in reducing test anxiety, and has great potential in benefiting all students in test and anxiety reduction, provided the person is not allergic to the oil. The use of lavender also appears to help sleep without the adverse effects of commonly used drugs Further, the anxiolytic effects of the oil might reduce unhealthy behaviors that students engage in, e.g. alcohol and drug use/overuse, to reduce stress and relax, and positively affect sleep.

ELIGIBILITY:
Inclusion Criteria:

* nursing students
* 18 years of age or older
* Male or Female
* all ethnicities will be included

Exclusion Criteria:

* cognitive impairments interring with reading, comprehending, following directions
* unstable psychiatric impairments
* chronic depression
* severe anxiety disorders
* asthma,
* fragrance allergy
* rhinitis
* upper respiratory tract infection
* lower respiratory tract infection
* smell/odor impairments
* allergies to plant-based essential oils
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Anxiety | From date of enrollment to up to 52 weeks
  Number of participants with anxiety
Test anxiety | From date of enrollment to up to 52 weeks
  Number of participants with test anxiety prior to examinations
Perceived stress | From date of enrollment to up to 52 weeks
  Number of participants who perceive stress before taking an examination
nausea or queasiness | From date of enrollment to up to 52 weeks
  Number of participants who have nausea and/or queasiness prior to examinations
Exam grade | From date of enrollment to up to 52 weeks
  Number of participants who take a specific course examination

SECONDARY OUTCOMES:
Grade point average (GPA) | From date of enrollment to up to 52 weeks
  Numerical indicator of cumulative grade success in the nursing program.

CONTACTS AND LOCATIONS:
Overall Officials: Martha J Greenberg, PhD, RN, Principal Investigator — Pace University

IPD SHARING:
Plan to Share IPD: No
I had not really considered it

REFERENCES:
- [Background] Hashemi N, Nazari F, Faghih A, Forughi M. Effects of blended aromatherapy using lavender and damask rose oils on the test anxiety of nursing students. J Educ Health Promot. 2021 Sep 30;10:349. doi: 10.4103/jehp.jehp_88_21. eCollection 2021. PMID 34761035
- [Background] Ozer Z, Teke N, Turan GB, Bahcecik AN. Effectiveness of lemon essential oil in reducing test anxiety in nursing students. Explore (NY). 2022 Sep-Oct;18(5):526-532. doi: 10.1016/j.explore.2022.02.003. Epub 2022 Feb 10. PMID 35190270
- [Background] Kaur Khaira M, Raja Gopal RL, Mohamed Saini S, Md Isa Z. Interventional Strategies to Reduce Test Anxiety among Nursing Students: A Systematic Review. Int J Environ Res Public Health. 2023 Jan 10;20(2):1233. doi: 10.3390/ijerph20021233. PMID 36673999
- [Background] Johnson CE. Effect of Inhaled Lemon Essential Oil on Cognitive Test Anxiety Among Nursing Students. Holist Nurs Pract. 2019 Mar/Apr;33(2):95-100. doi: 10.1097/HNP.0000000000000315. PMID 30747778